CLINICAL TRIAL: NCT06239272
Title: NRSTS2021, A Risk Adapted Study Evaluating Maintenance Pazopanib, Limited Margin, Dose-Escalated Radiation Therapy and Selinexor in Non-Rhabdomyosarcoma Soft Tissue Sarcoma (NRSTS)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NRSTS2021; NCI-2024-02554 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Adipocytic Neoplasm; Liposarcoma; Atypical Fibroxanthoma; Angiomatoid Fibrous Histiocytoma; Myoepithelioma; Fibrosarcoma NOS; Myxofibrosarcoma; Angiosarcoma; Osteosarcoma, Extraskeletal
Keywords: non-rhabdomyosarcoma; Proton therapy; Soft tissue sarcoma; Adipocytic Tumors; Fibroblastic/myofibroblastic Tumors; Dermatofibrosarcoma protuberans, fibrosarcomatous; Solitary fibrous tumor; Inflammatory myofibroblastic tumor; Low-grade myofibroblastic sarcoma; Superficial CD34-positive fibroblastic tumor; Myxoinflammatory fibroblastic sarcoma; Fibrohistiocytic Tumors; Plexiform fibrohistiocytic tumor; Giant cell tumor of soft parts NOS; Vascular Tumors; Pericytic Tumors; Smooth Muscle Tumors; Smooth muscle tumor of uncertain malignant potential; EBV-associated smooth muscle tumor; Ossifying fibromyxoid tumor; Undifferentiated Small Round Cell Sarcomas of Bone and Soft Tissue; Well differentiated liposarcoma: lipoma-like, sclerosing, inflammatory; Dedifferentiated liposarcoma; Myxoid Liposarcoma; Pleomorphic liposarcoma; Myxoid pleomorphic liposarcoma; Solitary fibrous tumor, malignant; Low grade fibromyxoid sarcoma; Sclerosing epithelioid fibrosarcoma; Malignant tenosynovial giant cell tumor; Epithelioid hemangioendothelioma; Glomus tumor; malignant; Inflammatory leiomyosarcoma; Malignant peripheral nerve sheath tumor; Melanotic malignant nerve sheath tumor; Granular cell tumor, malignant; Perineurioma, malignant; Phosphaturic mesenchymal tumor, malignant; NTRK-rearranged spindle cell neoplasm; Epithelioid sarcoma: proximal and classic variant; Clear cell sarcoma; Extraskeletal myxoid chondrosarcoma; Perivascular epithelioid tumor, malignant; Intimal sarcoma; Ossifying fibromyxoid tumor, malignant; Myoepithelial carcinoma; Undifferentiated sarcoma; Spindle cell sarcoma, undifferentiated; Pleomorphic sarcoma, undifferentiated; Round cell sarcoma, undifferentiated; Round cell sarcoma with EWSR1-non-ETS fusions; CIC-rearranged sarcomas; Sarcoma with BCOR genetic alteration
MeSH Terms: conditions — Neoplasms, Adipose Tissue; Liposarcoma; Histiocytoma, Angiomatoid Fibrous; Myoepithelioma; Fibrosarcoma; Dermatofibrosarcoma; Hemangiosarcoma; Osteosarcoma; Sarcoma; Granuloma, Plasma Cell; Solitary Fibrous Tumors; Vascular Neoplasms; Smooth Muscle Tumor; Liposarcoma, Myxoid; Hemangioendothelioma, Epithelioid; Glomus Tumor; Neurofibrosarcoma; Granular Cell Tumor; Nerve Sheath Neoplasms; Sarcoma, Clear Cell; Chondrosarcoma, Extraskeletal Myxoid; Disorders of Sex Development | interventions — Proton Therapy; pazopanib; Ifosfamide; Doxorubicin; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Low-Risk Subset A (Experimental): Participants with low grade tumors of any size, or high-grade tumors < 5 cm that have been (or are expected to be) completely removed by surgery. When the pathologist reviews the tumor specimen, the tissue around the tumor (margins) must be negative for cancer cells, meaning all of the cancer has been removed. These participants will have surgery to remove the tumor, followed by close observation. There will no further therapy after surgery, just monitoring for tumor recurrence and any side effects from surgery.
  Interventions: Procedure: Surgical resection; Radiation: Proton beam radiation therapy
- Low-Risk Subset B (Experimental): Participants with high-grade tumors that are < 5 cm with positive margins. This means that the pathologist finds cancer cells at the edge of the tissue, suggesting that all of the cancer has not been removed. These participants will have surgery followed by radiation therapy for about 5-6 weeks.
  Interventions: Procedure: Surgical resection; Radiation: Proton beam radiation therapy
- Intermediate-Risk Subset A (participants with low grade tumors): (Experimental): * If your tumor is completely removed at surgery [meaning the tissue around the tumor (margins) is negative for tumor cells], you will receive no further therapy and you will be closely observed for any signs of tumor recurrence.
  * If your tumor cannot be completely removed at surgery [meaning the tissue around the tumor (margins) is positive for tumor cells] and the tumor is low-grade, you will get consolidation therapy with additional chemotherapy and radiation therapy, followed by 6 months of maintenance therapy with pazopanib.
  Interventions: Procedure: Surgical resection; Radiation: Proton beam radiation therapy; Drug: Pazopanib; Drug: Ifosfamide; Drug: Doxorubicin
- Intermediate-Risk Subset B (participants with high-grade tumors between 5 and 10 cm in size (Experimental): * If your tumor is completely removed at surgery [meaning the tissue around the tumor (margins) is negative for tumor cells] you will continue with consolidation chemotherapy with additional chemotherapy without radiation therapy, followed by 6 months of maintenance therapy with pazopanib.
  * If your tumor cannot be completely removed at surgery [meaning the tissue around the tumor (margins) is positive for tumor cells], you will get consolidation therapy with additional chemotherapy and radiation therapy, followed by 6 months of maintenance therapy with pazopanib.
  Interventions: Procedure: Surgical resection; Radiation: Proton beam radiation therapy; Drug: Pazopanib; Drug: Ifosfamide; Drug: Doxorubicin
- Intermediate-Risk Subset C (participants with high-grade tumors > 10 cm): (Experimental): * After 3 cycles of induction chemotherapy, your doctor may decide to give an additional 4th cycle if he/she thinks it would be beneficial before surgery.
  * You will get consolidation therapy with additional chemotherapy and radiation therapy, followed by 6 months of maintenance therapy with pazopanib. The dose of radiation that you receive will be higher if your tumor cannot be completely removed at surgery (positive margins).
  Interventions: Procedure: Surgical resection; Radiation: Proton beam radiation therapy; Drug: Pazopanib; Drug: Ifosfamide; Drug: Doxorubicin
- High-Risk - 2 groups (Experimental): * If you have a low-grade tumor that has spread to other parts of the body AND the surgeon was able to completely remove all tumors from all parts of your body, you will have no further therapy after surgery. You will be closely followed to monitor you for any signs of tumor recurrence.
  * If you have a high-grade tumor OR a tumor that cannot be completely removed by surgery OR you have the CIC-DUX4 mutation, you will get consolidation chemotherapy and radiation therapy, followed by 6 months of maintenance therapy with pazopanib.
  Interventions: Procedure: Surgical resection; Radiation: Proton beam radiation therapy; Drug: Pazopanib; Drug: Ifosfamide; Drug: Doxorubicin; Drug: Selinexor

INTERVENTIONS:
Procedure: Surgical resection — Low, Intermediate and High-risk Surgery to remove tumor (standard of care)
Radiation: Proton beam radiation therapy — Low, Intermediate and High-risk Radiation therapy is considered standard of care for patients with NRSTS who have positive tumor margins. However, the dose that will be given in this study is higher than what is usually given, therefore, the dose of radiation in this study is research. Radiation will start about 3 to 6 weeks after your surgery, depending on how quickly you recover from surgery. Radiation will be given daily (Monday through Friday) for about 5 to 6 weeks.
Drug: Pazopanib — Intermediate and High-risk By mouth, either by tablet or a liquid suspension, 7 doses, days 1 to 7
  Other Names: VOTRIENT®
  Arms: High-Risk - 2 groups; Intermediate-Risk Subset A (participants with low grade tumors):; Intermediate-Risk Subset B (participants with high-grade tumors between 5 and 10 cm in size; Intermediate-Risk Subset C (participants with high-grade tumors > 10 cm):
Drug: Ifosfamide — Intermediate and High-risk Ifosfamide is a structural analogue of cyclophosphamide. Into the vein (IV) over about 3 hours, 3 doses, days 1, 2, and 3
  Other Names: Ifex
  Arms: High-Risk - 2 groups; Intermediate-Risk Subset A (participants with low grade tumors):; Intermediate-Risk Subset B (participants with high-grade tumors between 5 and 10 cm in size; Intermediate-Risk Subset C (participants with high-grade tumors > 10 cm):
Drug: Doxorubicin — Intermediate and High-risk An anthracycline antibiotic isolated from cultures of Streptomyces peucetius. Intermediate, High-risk Into the vein (IV) over about 1 hour, 2 doses, days 1 and 2
  Other Names: Adriamycin®; Rubex®
  Arms: High-Risk - 2 groups; Intermediate-Risk Subset A (participants with low grade tumors):; Intermediate-Risk Subset B (participants with high-grade tumors between 5 and 10 cm in size; Intermediate-Risk Subset C (participants with high-grade tumors > 10 cm):
Drug: Selinexor — High-risk Dosage and route of administration: Selinexor tablets for oral administration should be taken at approximately the same time each day without regards to meals.
  Selinexor is a selective inhibitor of nuclear export (SINE). Selinexor specifically blocks XPO1-mediated nuclear export by forming a slowly reversible covalent bond with the nuclear export protein XPO1 By mouth, either by tablet or a liquid suspension, 1 dose and day 3
  Other Names: XPOVIO®
  Arms: High-Risk - 2 groups

SUMMARY:
The study participant has been diagnosed with non-rhabdomyosarcoma (NRSTS).

Primary Objectives

Intermediate-Risk

* To estimate the 3-year event-free survival for intermediate-risk patients treated with ifosfamide, doxorubicin, pazopanib, surgery, and maintenance pazopanib, with or without RT.
* To characterize the pharmacokinetics of pazopanib and doxorubicin in combination with ifosfamide in intermediate-risk participants, to assess potential covariates to explain the inter- and intra-individual pharmacokinetic variability, and to explore associations between clinical effects and pazopanib and doxorubicin pharmacokinetics.

High-Risk

* To estimate the maximum tolerated dose (MTD) and/or the recommended phase 2 dosage (RP2D) of selinexor in combination with ifosfamide, doxorubicin, pazopanib, and maintenance pazopanib in high-risk participants.
* To characterize the pharmacokinetics of selinexor, pazopanib and doxorubicin in combination with ifosfamide in high-risk participants, to assess potential covariates to explain the inter- and intra-individual pharmacokinetic variability, and to explore associations between clinical effects and selinexor, pazopanib and doxorubicin pharmacokinetics.

Secondary Objectives

* To estimate the cumulative incidence of primary site local failure and distant metastasis-free, disease-free, event-free, and overall survival in participants treated on the risk-based treatment strategy defined in this protocol.
* To define and describe the CTCAE Grade 3 or higher toxicities, and specific grade 1-2 toxicities, in low- and intermediate-risk participants.
* To study the association between radiation dosimetry in participants receiving radiation therapy and the incidence and type of dosimetric local failure, normal adjacent tissue exposure, and musculoskeletal toxicity.
* To evaluate the objective response rate (complete and partial response) after 3 cycles for high-risk patients receiving the combination of selinexor with ifosfamide, doxorubicin, pazopanib, and maintenance pazopanib.
* To assess the relationship between the pharmacogenetic variation in drug-metabolizing enzymes or drug transporters and the pharmacokinetics of selinexor, pazopanib, and doxorubicin in intermediate- or high-risk patients.

Exploratory Objectives

* To explore the correlation between radiographic response, pathologic response, survival, and toxicity, and tumor molecular characteristics, as assessed through next-generation sequencing (NGS), including whole genome sequencing (WGS), whole exome sequencing (WES), and RNA sequencing (RNAseq).
* To explore the feasibility of determining DNA mutational signatures and homologous repair deficiency status in primary tumor samples and to explore the correlation between these molecular findings and the radiographic response, survival, and toxicity of patients treated on this protocol.
* To explore the feasibility of obtaining DNA methylation profiling on pretreatment, post-induction chemotherapy, and recurrent (if possible) tumor material, and to assess the correlation with this and pathologic diagnosis, tumor control, and survival outcomes where feasible.
* To explore the feasibility of obtaining high resolution single-cell RNA sequencing of pretreatment, post-induction chemotherapy, and recurrent (if possible) tumor material, and to characterize the longitudinal changes in tumor heterogeneity and tumor microenvironment.
* To explore the feasibility of identifying characteristic alterations in non-rhabdomyosarcoma soft tissue sarcoma in cell-free DNA (cfDNA) in blood as a non-invasive method of detecting and tracking changes during therapy, and to assess the correlation of cfDNA and mutations in tumor samples.
* To describe cardiovascular and musculoskeletal health, cardiopulmonary fitness among children and young adults with NRSTS treated on this protocol.
* To investigate the potential prognostic value of serum cardiac biomarkers (high-sensitivity cardiac troponin I (hs-cTnI), N-terminal pro B-type natriuretic peptide (NT-Pro-BNP), serial electrocardiograms (EKGs), and serial echocardiograms in patients receiving ifosfamide, doxorubicin, and pazopanib, with or without selinexor.
* To define the rates of near-complete pathologic response (>90% necrosis) and change in FDG PET maximum standard uptake value (SUVmax) from baseline to week 13 in intermediate risk patients with initially unresectable tumors treated with induction pazopanib, ifosfamide, and doxorubicin, and to correlate this change with tumor control and survival outcomes.
* To determine the number of high-risk patients initially judged unresectable at diagnosis that are able to undergo primary tumor resection after treatment with ifosfamide, doxorubicin, selinexor, and pazopanib.
* To identify the frequency with which assessment of volumes of interest (VOIs) of target lesions would alter RECIST response assessment compared with standard linear measurements.

DETAILED DESCRIPTION:
For the intermediate-risk group, a two-sided one-sample log-rank test will be used to detect an improvement in 3-year EFS from 72% to 86% (power 87% with type I error rate of 5%). With this design, 53 evaluable patients in total will be required. Non-binding interim futility rules will be employed for the combination of subsets of A, B, C at week 10 and a separate rule for subset B at year 2 in terms of local failure rate.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - All Patients

* Patients must be ≤ 30 years at the time of the biopsy that established the diagnosis of NRSTS.
* Surgical Resection: Patients who had an upfront resection prior to enrollment will be eligible if they are able to begin therapy within 28 days of resection assuming other eligibility criteria are met. Delayed resection is preferred for all patients with intermediate and high-risk disease.
* Lansky performance status score ≥ 60 for patients ≤ 16 years of age. Karnofsky performance status score ≥ 60 for patients >16 years of age. Note patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Diagnosis

• Patients with CIC-DUX 4 rearranged sarcomas will be enrolled on the high-risk stratum only, regardless of presence of metastasis, size, or resection status.

Patient has low-risk disease if the patient has a:

* Low-grade tumor of any size where R0 or R1 surgical margins are anticipated or achieved.
* High-grade tumors that are < 5 cm where R0 or R1 resection margins are anticipated or achieved.

Patient must have adequate organ function in the organs that will be within the radiotherapy field.

Adequate renal function defined as:

* Creatinine clearance or radioisotope GFR > 70 mL/min/1.73 m2, or
* A normal serum creatinine based on age/gender as follows

Age Maximum Serum Creatinine (mg/dL) Male Female 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4 > 16 years 1.5 1.4

Adequate liver function defined as:

* Total bilirubin < 1.5 x upper limit of normal (ULN) for age
* SGOT (AST) or SGPT (ALT) < 2.5 x ULN for age

Adequate cardiac function defined as:

* Ejection fraction of > 55% by echocardiogram or cardiac MRI
* QTc < 480 msec

Adequate pulmonary function defined as:

* No evidence of dyspnea at rest, no exercise intolerance, and a resting pulse oximetry reading > 94% on room air if there is clinical indication for determination.

Inclusion Criteria - Intermediate and High Risk Participants

Patient has intermediate-risk if the patient has a:

* Low-grade non-metastatic initially unresectable disease at study enrollment where delayed resection is planned.
* High-grade < 5 cm non-metastatic initially unresectable disease at study enrollment where delayed resection is planned. Of note, patients enrolled on the low-risk arm who were unable to achieve gross total resection where delayed re-resection is planned are eligible for this arm.
* High-grade tumor > 5 cm that is potentially resectable.

Patient high-risk if the patient has:

* Metastatic disease at presentation
* Unresectable disease at study enrollment where delayed resection is not anticipated. Of note, patients enrolled on the low-risk arm who were unable to achieve gross total resection where delayed re-resection is not-planned are eligible for this arm.
* CIC-DUX4 rearranged sarcoma

Organ Function

Adequate bone marrow function defined as:

* Absolute neutrophil count > 1000/µL
* Platelet count > 100,000/µL
* Hemoglobin > 8 g/dL for patients < 16 years of age
* Hemoglobin > 9 g/dL for patients > 16 years of age

Note: No transfusions are permitted 7 days prior to laboratory studies to determine eligibility.

Adequate renal function defined as:

* Creatinine clearance or radioisotope GFR > 70 mL/min/1.73 m2, or
* A normal serum creatinine based on age/gender as follows

Age Maximum Serum Creatinine (mg/dL) Male Female 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4 > 16 years 1.5 1.4

Adequate liver function defined as:

* Total bilirubin < 1.5 x upper limit of normal (ULN) for age
* SGOT (AST) or SGPT (ALT) < 2.5 x ULN for age

Adequate cardiac function defined as:

* Ejection fraction of > 55% by echocardiogram or cardiac MRI
* QTc < 480 msec

Adequate pulmonary function defined as:

* No evidence of dyspnea at rest, no exercise intolerance, and a resting pulse oximetry reading > 94% on room air if there is clinical indication for determination.

Anticoagulation

Patients on low molecular weight heparin, warfarin (with a stable INR), or direct oral anticoagulants (DOAC) who have been on a stable dose of are eligible. Patients being treated for a pulmonary embolism or deep venous thrombosis (DVT) must have been treated for a minimum of 6 weeks prior to starting therapy treatment.

Life Expectancy

Patient must have a life expectancy of at least 3 months with appropriate therapy.

Exclusion Criteria:

* Patients with known primary CNS sarcoma or CNS metastases are not eligible. Note: Brain imaging is not an eligibility requirement. Tumors with intracranial extension will be allowed.
* Patients with the following histologic diagnosis are not eligible: intermediate locally aggressive tumors as defined by WHO, malignant rhabdoid tumor, alveolar soft part sarcoma, infantile fibrosarcoma, unresectable/metastatic dermatofibrosarcoma protuberans, inflammatory myofibroblastic tumor, desmoid fibromatosis, rhabdomyosarcoma, desmoplastic small round cell tumor, BCOR-CCNB3 fusion positive sarcoma.
* Bleeding diathesis: Patients with evidence of active bleeding or bleeding diathesis will be excluded (Note: Patients aged > 17 years with excess of 2.5 mL of hemoptysis are not eligible).
* Uncontrolled hypertension: Patients with uncontrolled hypertension (CTCAE v5 Grade ≥ 2) are ineligible. Hypertension must be well controlled on stable doses of medication for at least two weeks.

Prior Therapy

* Patients must have had no prior systemic therapy for the treatment of the NRSTS
* Patients must have had no prior anthracycline or ifosfamide chemotherapy
* Patients must have had no prior use of pazopanib or similar multi-targeted TKI.

Patients must have had no prior radiotherapy to tumor-involved sites.

Note: Patients previously treated for a non-NRSTS cancer are eligible provided they meet the prior therapy requirements. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier are excluded.

* CYP3A4 Substrates WITH Narrow Therapeutic Indices: Patients chronically receiving medications known to be metabolized by CYP3A4 and with narrow therapeutic indices within 7 days prior to study enrollment, including but not limited to pimozide, aripiprazole, triazolam, ergotamine and halofantrine are not eligible. Note: the use of fentanyl is permitted.
* CYP3A4 Inhibitors: Patients chronically receiving drugs that are known potent CYP3A4 inhibitors within 7 days prior to study enrollment, including but not limited to itraconazole, clarithromycin, erythromycin, many NNRTIs, diltiazem, verapamil, and grapefruit juice are not eligible.
* CYP3A4 Inducers: Patients chronically receiving drugs that are known potent CYP3A4 inducers within 14 days prior to study enrollment, including but not limited to carbamazepine, phenobarbital, phenytoin, rifampin, and St. John's wort are not eligible (with the exception of glucocorticoids).
* Certain medications that are associated with a risk for QTc prolongation and/or Torsade's de Pointes, although not prohibited, should be avoided or replaced with medications that do not carry these risks, if possible.
* Subjects with any condition that may impair the ability to absorb oral medications/investigational product including:

  * prior surgical procedures affecting absorption including, but not limited to major resection of stomach or small bowel
  * active peptic ulcer disease
  * malabsorption syndrome

3.4.12 Thyroid Replacement Therapy: Patients who require thyroid replacement therapy are not eligible if they have not been receiving a stable replacement dose for at least 4 weeks prior to study enrollment.

3.4.13 Subjects with any condition that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, including:

* active peptic ulcer disease
* known intraluminal metastatic lesions
* inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other gastrointestinal conditions which increase the risk of perforation
* history of abdominal fistula, gastrointestinal perforation or intra- abdominal abscess within 28 days prior to beginning study treatment.

3.4.14 Pulmonary embolism or DVT. Patients must not have experienced:

* An untreated pulmonary embolism or DVT in last 6 months or
* treated pulmonary embolism or DVT which has been treated with therapeutic anticoagulation for less than 6 weeks
* arterial thrombosis in last 12 months

History of serious or non-healing wound, ulcer, or bone fracture.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pazopanib. In addition, these subjects are at increased risk of lethal infections when treated with marrow-suppressive therapy.

Patients who are receiving any other investigational agent(s).

Pregnancy and Breast Feeding

* Pregnancy and Breast Feeding Female patients who are pregnant are ineligible due to risks of fetal and teratogenic adverse events as seen in animal/human studies.
* Lactating females are not eligible unless they have agreed not to breastfeed their infants during treatment and for a period of 1 month following completion of treatment.
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained.
* Unwillingness to use an effective contraceptive method for the duration of their study participation and for at least 1 month after treatment is completed if sexually active with reproductive potential.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 139 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2034-06 (Estimated); Study Completion 2037-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 9 years (6 years of accrual and 3 year follow-up after enrollment of last patient
  We will estimate the 3-year event-free survival for intermediate-risk patients, which is the estimated probability of a patient not having any events within the 3-year follow-up. The events are defined as including local failure, regional failure, distant failure, a subsequent malignant neoplasm, or death, whichever occurred first.
Maximum tolerated dose (MTD) and/or the recommended phase 2 dosage (RP2D) | 4 years]
  MTD is defined in the study as the highest treatment dose that would deliver desirable treatment effects without resulting in a target toxicity rate greater than 0.3. We will employ the Bayesian optimal interval (BOIN) design to find the MTD in high-risk participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gartrell, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (6):
- United States (6):
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Our Lady of the Lake Children's Hospital, Baton Rouge, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University Medical Center, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: SAP, ICF, CSR
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols